CLINICAL TRIAL: NCT02374814
Title: Immunogenicity of a Two vs Three Dose, Intradermal (ID) vs Intramuscular (IM) Administration of a Licensed Rabies Vaccine for Pre-Exposure Vaccination
Brief Title: Immunogenicity of Rabies Vaccine for Pre Exposure Prophylaxis
Acronym: RABVAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Timothy Endy, MD MPH, Chair, Microbiology and Immunology, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 568085
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Results first posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rabies vaccine IM 3 dose (Active Comparator): Intramuscular injection: 1mL at 0, 7 and 21 days. An additional 1 mL intramuscular dose at day 365
  Interventions: Drug: Rabies vaccine
- Rabies vaccine ID 3 dose (Experimental): Intradermal injection: 0.1mL at 0, 7 and 21 days. A single intramuscular 1 mL dose at day 365
  Interventions: Drug: Rabies vaccine
- Rabies vaccine IM 2 dose (Experimental): Intramuscular injection: 1mL at 0, 7 days. An additional 1 mL intramuscular dose at day 365
  Interventions: Drug: Rabies vaccine
- Rabies vaccine ID 2 dose (Experimental): Intradermal injection: 0.1mL at 0, 7 days. A single intramuscular 1 mL dose at day 365
  Interventions: Drug: Rabies vaccine
- Placebo IM 1 dose (Placebo Comparator): Albumin and saline comparator, Intramuscular injection: 1mL
  Interventions: Drug: Placebo
- Placebo ID 1 dose (Placebo Comparator): Albumin and saline comparator, Intradermal injection: 0.1mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rabies vaccine — Compare dose schedule and route of administration
  Other Names: Rabavert
  Arms: Rabies vaccine ID 2 dose; Rabies vaccine ID 3 dose; Rabies vaccine IM 2 dose; Rabies vaccine IM 3 dose
Drug: Placebo — Placebo
  Other Names: Albumin
  Arms: Placebo ID 1 dose; Placebo IM 1 dose

SUMMARY:
The purpose of this study is to compare the effectiveness of a two dose versus a three dose schedule and intramuscular versus intradermal injection for pre-exposure prophylaxis.

DETAILED DESCRIPTION:
This is an exploratory vaccine trial to evaluate immunogenicity of a non-licensed dosing schedule and route of administration for a currently FDA licensed rabies vaccine for pre-exposure prophylaxis against rabies infection. The goal of this study is to characterize the immune response and persistence of immunity to a shortened dose schedule and intradermal (ID) administration, relative to the current licensed dosing schedule of the rabies vaccine (3 dose (0, 7, 21 days) IM). Rabies virus is endemic throughout the world due to high rates of both wild and domestic animal rabies and the risk to deployed military in endemic areas is considerable. Currently the commonly supported pre-exposure prophylaxis regimen for rabies, in the United States is comprised of three, 1.0 ml intramuscular (IM) injections of the human diploid cell vaccine (HDCV) or purified chick embryo cell (PCEC) rabies vaccine on days 0, 7, and 21 or 28. Modified, two and three dose schedules of intradermal (ID) injections of 0.1 ml of HDCV and PCEC are utilized outside the US. These two and three dose intradermal schedules share a similar safety and immunogenicity profile to intramuscular vaccinations and are easily boosted at one year after vaccination. A death, from rabies, of a US Soldier returned from Afghanistan underscores the importance of rabies pre-exposure prophylaxis for soldiers and the need to evaluate the safest, most effective means of vaccinating large deploying forces. While the current three dose, 1 ml IM rabies series is effective, a shortened, equally effective vaccination series with significantly smaller dose per injection would greatly improve the logistics and cost associated with universal or even targeted coverage of deploying soldiers. Evaluation of a shorter, smaller-dose, pre-exposure vaccination series for rabies is the goal of this study.

ELIGIBILITY:
Inclusion Criteria:

Male and non-pregnant females aged ≥ 18 to ≤ 60 years on the day of inclusion Able to comprehend and give informed consent Able to attend all scheduled visits and to comply with all trial procedures Subject in good health, based on medical history and physical examination

Exclusion Criteria:

1. Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post- menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
2. Participation in the 4 weeks preceding the first trial vaccination, or planned participation during the present trial period, in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
3. Previous history of receiving the rabies vaccine.
4. Previous history of receiving rabies immune globulin.
5. Any major psychiatric disorder, such as severe depression, severe anxiety disorder, psychosis, schizophrenia, other major psychiatric disorders, or seizures. History of mild depression or anxiety disorder that is well controlled is not an exclusion criteria.
6. Any history of cardiac arrhythmias, such as: Bradycardia, tachycardia, heart block, SVT, PAC, VF, VT, or any other conduction abnormalities.
7. Use of any immunosuppressive drug , including topical steroids of potency groups I, II or III within 30 days of the study period.
8. Any immunosuppressive disorder, such as HIV, common variable, active cancers or chemotherapy.
9. History of renal insufficiency or requiring dialysis.
10. Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
11. Identified as an employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employee or the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polhemus, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- State University of New York, Upstate Medical University (SUNY-UMU), Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Endy TP, Keiser PB, Wang D, Jarman RG, Cibula D, Fang H, Ware L, Abbott M, Thomas SJ, Polhemus ME. Serologic Response of 2 Versus 3 Doses and Intradermal Versus Intramuscular Administration of a Licensed Rabies Vaccine for Preexposure Prophylaxis. J Infect Dis. 2020 Apr 7;221(9):1494-1498. doi: 10.1093/infdis/jiz645. PMID 31802120

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject in group 4 was lost to follow up prior to receiving vaccine.
Groups:
- Rabies Vaccine IM 3 Dose: Rabies vaccine: 1.0 ml delivered Intramuscularly (IM) on day 0, 7, 21 and 365.
- Rabies Vaccine ID 3 Dose: Rabies vaccine: 0.1 ml of rabies vaccine delivered intradermal (ID) on days 0, 7, and 21 with a 1.0ml boost delivered IM on day 365.
- Rabies Vaccine IM 2 Dose: Rabies vaccine: 1.0ml delivered IM on day 0, 7 and 365.
- Rabies Vaccine ID 2 Dose: Rabies vaccine: 0.1ml delivered on day 0 and 7 with a 1.0ml IM boost on day 365
- Placebo IM 1 Dose: Placebo: 1.0ml delivered IM on day 0
- Placebo ID 1 Dose: Placebo: 0.1ml delivered on day 0
Period: Overall Study
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose
Started | 12 | 12 | 12 | 11 | 6 | 6
Completed | 11 | 11 | 11 | 9 | 6 | 6
Not Completed | 1 | 1 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who received at least one dose of rabies vaccine or placebo
Groups:
- Rabies Vaccine IM 3 Dose: This is standard FDA approved schedule
  Rabies vaccine: Compare dose schedule and route of administration
- Rabies Vaccine ID 3 Dose: This is using alternative administration method
  Rabies vaccine: Compare dose schedule and route of administration
- Rabies Vaccine IM 2 Dose: This is using alternative dose schedule
  Rabies vaccine: Compare dose schedule and route of administration
- Rabies Vaccine ID 2 Dose: This is using alternative dose schedule and administration
  Rabies vaccine: Compare dose schedule and route of administration
- Placebo IM 1 Dose; Placebo ID 1 Dose: Albumin and saline comparator
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose | Total
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 6 | 6 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 12 | 12 | 12 | 10 | 6 | 6 | 58
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (7.0) | 29.3 (9.5) | 32.3 (10.0) | 31.8 (12.6) | 38.5 (15.3) | 35.7 (10.6) | 32.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 8 | 4 | 3 | 38
  Male | 5 | 4 | 4 | 3 | 2 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 12 | 12 | 11 | 6 | 4 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 0 | 0 | 3
  White | 12 | 9 | 10 | 11 | 6 | 6 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 11 | 6 | 6 | 59

OUTCOME MEASURES:

1. Primary Outcome: Protective Humoral Immune Response at 1 Month Post First Vaccination.
Description: Percentage of subjects achieving the protective titer of ≥ 0.5 IU/ml against rabies virus
Time Frame: 1 month post first vaccination
Population: Placebo groups were used for adverse event data collection only. It was not expected that placebo group would elicit any antibody titer to rabies. Samples in groups 5 and 6 were not analyzed for primary or secondary outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Rabies Vaccine IM 3 Dose: Rabies vaccine:
  Intramuscular injection: 1mL at 0, 7 and 21 days. An additional 1 mL intramuscular dose at day 365.
- Rabies Vaccine ID 3 Dose: Rabies vaccine:
  Intradermal injection: 0.1mL at 0, 7 and 21 days. A single intramuscular 1 mL dose at day 365.
- Rabies Vaccine IM 2 Dose: Rabies vaccine:
  Intramuscular injection: 1mL at 0, 7 days. An additional 1 mL intramuscular dose at day 365.
- Rabies Vaccine ID 2 Dose: Rabies vaccine:
  Intradermal injection: 0.1mL at 0, 7 days. A single intramuscular 1 mL dose at day 365.
- Placebo IM 1 Dose: Albumin and saline comparator
  Placebo: A single 1mL intramuscular injection at day 0
- Placebo ID 1 Dose: Albumin and saline comparator
  Placebo: A single intradermal injection of 0.1mL at day 0
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 0 | 0
Participants | 12 | 12 | 12 | 11 |  |

2. Primary Outcome: Protective Humoral Immune Response 12 Months Post First Vaccination.
Description: Percentage of subjects achieving the protective titer of ≥ 0.5 IU/ml against rabies virus 12 months post vaccinations (prior to boost).
Time Frame: 12 months post first vaccination
Population: One subject in each of groups 1, 2, and 4 were lost to follow up prior to vaccination boost. Placebo groups were used for adverse event data collection only. It was not expected that placebo group would elicit any antibody titer to rabies. Samples in groups 5 and 6 were not analyzed for primary or secondary outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo ID 1 Dose: Albumin and saline comparator
  Placebo: A single 0.1mL intradermal injection at day 0
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose
Number analyzed (Participants) | 11 | 11 | 12 | 10 | 0 | 0
Participants | 7 | 5 | 7 | 6 |  |

3. Secondary Outcome: Protective Humoral Immune Response 7 Days Post Booster at 12 Months Post First Vaccination.
Description: Percentage of subjects achieving the protective titer of ≥ 0.5 IU/ml against rabies virus at 7 days post boost.
Time Frame: up to 13 months post first vaccination
Population: One subject in group 3 and one in 4 withdrew consent not due to adverse events. Placebo groups were used for adverse event data collection only. It was not expected that placebo group would elicit any antibody titer to rabies. Samples in groups 5 and 6 were not analyzed for primary or secondary outcome measures.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo IM 1 Dose: Albumin and saline comparator
  Placebo: 1mL intramuscular at day 0
- Placebo ID 1 Dose: Albumin and saline comparator
  Placebo: 0.1 mL intradermal at day 0
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose
Number analyzed (Participants) | 11 | 11 | 11 | 9 | 0 | 0
Participants | 11 | 11 | 11 | 9 |  |

ADVERSE EVENTS:
Time Frame: 372 days for all groups (1-4) receiving rabies vaccine; 7 days for groups 5-6 receiving control
Groups:
- Placebo IM 1 Dose: Albumin and saline comparator
  Intramuscular injection: 1ml
- Placebo ID 1 Dose: Albumin and saline comparator
  Intradermal injection: 0.1ml
Arm/Group | Rabies Vaccine IM 3 Dose | Rabies Vaccine ID 3 Dose | Rabies Vaccine IM 2 Dose | Rabies Vaccine ID 2 Dose | Placebo IM 1 Dose | Placebo ID 1 Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/11 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/11 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 10/12 | 12/12 | 8/12 | 11/11 | 1/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabies Vaccine IM 3 Dose (N=12) | Rabies Vaccine ID 3 Dose (N=12) | Rabies Vaccine IM 2 Dose (N=12) | Rabies Vaccine ID 2 Dose (N=11) | Placebo IM 1 Dose (N=6) | Placebo ID 1 Dose (N=6)
Injection site reaction (General disorders) | 7 | 11 | 6 | 10 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 1 | 0 | 0
Flu-like symptoms (General disorders) | 2 | 0 | 1 | 3 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Fever (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT02374814/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT02374814/SAP_001.pdf
  • Informed Consent Form (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT02374814/ICF_002.pdf